CLINICAL TRIAL: NCT05555251
Title: Phase 1/2a Open-label Clinical Trial of BI-1607, an Fc-Engineered Monoclonal Antibody to CD32b (FcγRIIB), in Combination with Trastuzumab in Subjects with HER2-positive Advanced Solid Tumors
Brief Title: BI-1607 in Combination with Trastuzumab in Subjects with HER2-positive Advanced Solid Tumors
Acronym: CONTRAST
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After the completion of phase IA, for business reasons it was decided to terminate the study.
Sponsor: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-BI-1607-01
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Metastatic Breast Cancer; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Gastric Adenocarcinoma
Keywords: HER2-positive; solid tumours
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2a, FIH, open-label, multicenter, dose-escalation, consecutive-cohort study of BI-1607 in combination with trastuzumab.
  The study will consist of 2 Phases:
  * Phase 1, the dose-escalation part of the study, the aim of which is to assess safety and tolerability and to determine the RP2D of BI-1607 in combination with trastuzumab in subjects with HER2+ advanced solid tumors.
  * Phase 2a, comprising of 2 separate expansion cohorts treated at the RP2D of BI-1607 in combination with trastuzumab in subjects with locally advanced or metastatic HER2+ breast cancer and subjects with HER2+ metastatic gastric or gastroesophageal junction adenocarcinoma. The aim of Phase 2a is to collect additional safety data to further support RP2D, and to detect early signs of clinical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I -Dose escalation (Experimental): Dose escalation study of BI-1607 combined with trastuzumab in HER2+ advanced or metastatic solid tumors.
  Interventions: Drug: BI-1607; Drug: Trastuzumab
- Phase 2a - Expansion cohorts (Experimental): Dose expansion study of BI-1607 combined with trastuzumab in cohort 1: HER2 positive locally advanced or metastatic HER2+ breast cancer and cohort 2: metastatic gastric or gastroesophageal junction adenocarcinoma
  Interventions: Drug: BI-1607; Drug: Trastuzumab

INTERVENTIONS:
Drug: BI-1607 — administered at different doses in Phase I by intravenous infusions every 3 weeks.
  Arms: Phase I -Dose escalation
Drug: BI-1607 — administered at the recommended dose in Phase 2a by intravenous infusions every 3 weeks.
  Arms: Phase 2a - Expansion cohorts
Drug: Trastuzumab — administered at 8mg/kg for the first infusion and at 6mg/kg in subsequent infusions by intravenous infusions every 3 weeks.
  Other Names: Herceptin

SUMMARY:
HER2+ breast and gastric cancer patients' survival is significantly improved by trastuzumab alone or in combination with chemotherapy. However, many patients remain uncured and develop resistance to trastuzumab resulting in relapse or progression of the disease. BI-1607, a human immunoglobulin G1 (IgG1) monoclonal antibody (mAb) targets CD32b (Fc Gamma Receptor IIB), it is intended to enhance the efficacy and overcome resistance to existing cancer treatments such as trastuzumab.

This is a Phase 1/2a, first-in-human, open-label, multicenter, dose-escalation, consecutive-cohort study of BI-1607 in combination with trastuzumab in subjects with HER2+ advanced solid tumors whose tumor has progressed after standard therapy.

DETAILED DESCRIPTION:
This is a Phase 1/2a, first-in-human, open-label, multicenter, dose-escalation, consecutive-cohort study of BI-1607 in combination with trastuzumab in subjects with HER2+ advanced solid tumors whose tumor has progressed after standard therapy.

The Phase 1 part of the trial is a dose escalation study of BI-1607 combined with trastuzumab in HER2+ advanced or metastatic solid tumors, the aim is to assess safety and tolerability and to determine the recommended phase II dose of BI-1607 in combination with trastuzumab.

The selected dose of BI-1607 will be studied in a subsequent Phase 2a part of the trial along with trastuzumab in 2 open-label, expansion cohorts of 15 evaluable subjects each. The first cohort will enroll subjects with locally advanced or metastatic HER2+ breast cancer, and the second will recruit subjects with HER2+ metastatic gastric or gastroesophageal junction adenocarcinoma. The aim of the phase 2a is to collect additional safety data to further support the recommended dose, and to detect early signs of clinical activity.

ELIGIBILITY:
Main Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial.
* Is ≥18 years of age on day of signing informed consent.
* Has received standard of care or is intolerant to standard of care antineoplastic therapy. Subjects who are intolerant to trastuzumab cannot be enrolled in the study.
* Has at least 1 measurable disease lesion as defined by RECIST v1.1 criteria.
* Has a locally confirmed HER2+ tumor.
* Must have progressive disease after the last line of treatment. In addition, subjects must have received the following previous lines of treatment:

  1. Prior lines of treatment including trastuzumab and chemotherapy.
  2. At least one prior line of treatment with an antibody-drug conjugate (ADC) (eg, trastuzumab-emtansine [TDM-1, or trastuzumab-deruxtecan]).

Main Exclusion Criteria:

* Needs doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) while on the trial other than as premedication.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has cardiac or renal amyloid light-chain amyloidosis.
* Has had clinically significant lung disease requiring systemic corticosteroid treatment within the last 6 months of enrollment.
* Has an active, known, or suspected autoimmune disease.
* Is at high medical risk because of nonmalignant systemic disease including severe active infections on treatment with antibiotics, antifungals, or antivirals.
* Has presence of chronic graft versus host disease.
* Has had an allogenic tissue/solid organ transplant.
* Has uncontrolled or significant cardiovascular disease.
* Has a known additional malignancy of another type, except for adequately treated cone-biopsied carcinoma in situ (eg, breast carcinoma, cervical cancer in situ), adequately controlled superficial bladder cancer, and basal or squamous cell carcinoma of the skin.
* Has a diagnosis of primary or acquired immunodeficiency disorder or is taking any other form of immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability profile of BI-1607 in combination with trastuzumab | End of treatment visit or 30 days after last dose of study drug.
  Adverse events (AEs) and serious adverse events (SAEs) (graded according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v5.0) and their causality in relation to BI-1607 or to the combination with trastuzumab
Identify Dose limiting toxicities, determine the maximum tolerate dose of BI-1607 and propose a recommended Phase 2 dose (RP2D) for evaluation of BI-1607 in combination with trastuzumab. | 22 days
  Occurrence of DLTs

SECONDARY OUTCOMES:
Assessment of the pharmacokinetic (PK) profile of BI-1607 when administered every 3 weeks in combination with trastuzumab | 90 days after the last dose of BI-1607
  The PK parameters will include area under the serum concentration-time curve, maximum concentration, time to maximum concentration, and terminal half-life
Assessment of the immunogenicity of BI-1607 when administered in combination with trastuzumab | 90 days after the last dose of BI-1607
  Antidrug antibody response to BI-1607 in blood serum
Assessment of the CD32b receptor occupancy (RO) of BI-1607 on B cells when administered in combination with trastuzumab | 30 days after the last dose of BI-1607
  RO on circulating B lymphocytes
Assessment of the possible antitumor activity of BI-1607 in combination with trastuzumab | 1 year after the last treatment
  Best tumor response, objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, progression-free survival (PFS), time to response, duration of response (DOR) and OS

OTHER OUTCOMES:
Exploratory: investigate expression levels of Fc receptors, and other immunological markers on immune cells infiltrating the tumor | 1 day
  Expression levels of Fc receptors (eg, CD32b) and other markers of immunological activity using immunohistochemistry (IHC) and/or nucleotide-based assays using tissue samples
Exploratory: investigate the genetic background of subjects with respect to FcgammaR isoforms and explore a potential correlation of the genetic background with clinical responses | 1 day
  Determination of Fcgamma receptor isoforms using nucleotide-based assays on genetic material extracted from whole blood
Exploratory: explore any exposure-response and/or exposure-safety relationship between BI-1607 serum concentrations and clinical outcome | 1 day
  Correlation of BI-1607 PK and antitumor activity measures, as well as to safety measures of interest

CONTACTS AND LOCATIONS:
Overall Officials: Andres McAllister, MD, PhD, Study Director — BioInvent International AB
Locations (6):
- Germany (2):
  - Evang. Kliniken Essen-Mitte, Essen
  - Krankenhaus Nordwest, Frankfurt
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Complejo hospitalario Ruber Juan Bravo, Madrid
- United Kingdom (2):
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Cortes J, Priego A, Garralda E, Rojas K, Lord SR, Goetze TO, Kuemmel S, Crabb SJ, Parra-Guillen ZP, Borggren M, Karlsson I, Lindahl D, Martensson L, Oldham R, Ropenga A, Teige I, Wallin J, Frendeus B, McAllister A. A First-in-Class mAb (BI-1607) Targeting FcgammaRIIB: Preclinical Data and First-in-Human Studies in Patients with HER2-Positive Advanced Solid Tumors. Clin Cancer Res. 2025 Dec 1;31(23):4953-4963. doi: 10.1158/1078-0432.CCR-25-1348. PMID 41071338